CLINICAL TRIAL: NCT03724929
Title: Value of Pharmacokinetic Assays (Vedolizumab and Anti-vedolizumab Antibody) in the Prediction of Induction and Maintenance Therapeutic Response in Ulcerative Colitis
Brief Title: Value of Pharmacokinetic Assays in the Prediction of Therapeutic Response in Ulcerative Colitis
Acronym: PREDIRESPUC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to lack of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Takeda (Industry); Theradiag (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1708213; 2018-001051-12 (EudraCT Number)
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Vedolizumab; anti-vedolizumab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ulcerative Colitis patients (Experimental): To determine if the best cut-off points of vedolizumab (VDZ) trough levels measured at W6 capable to identify UC patients who will achieve a clinical response at week 10 with VDZ and also the best cut-off points of VDZ trough levels measured at W14 capable to identify UC patients who will achieve a clinical remission to maintenance therapy with VDZ :
  Blood samples will be systematically collected at W0, W2, W6, W14 and W52 for vedolizumab pharmacokinetic parameters, including the vedolizumab trough levels and the specific anti-vedolizumab antibody. A supplementary blood sample will be collected at W10 which is the point where a significant greater number of patients were in remission.
  Rectosigmoidoscopy will be performed in each center at time points W0, W10 and W52, to evaluate treatment efficacy.
  In cases of loss of response, rectosigmoidoscopy will be performed before and four weeks after optimization.
  Interventions: Procedure: Blood sample; Device: Rectosigmoidoscopy

INTERVENTIONS:
Procedure: Blood sample — Blood samples will be systematically collected at W0, W2, W6, W14 and W52 for vedolizumab pharmacokinetic parameters, including the vedolizumab trough levels and the specific anti-vedolizumab antibody. A supplementary blood sample will be collected at W10 which is the point where a significant greater number of patients were in remission.
Device: Rectosigmoidoscopy — Rectosigmoidoscopy will be performed in each center at time points W0, W10 and W52.

SUMMARY:
Vedolizumab (VDZ) is a monoclonal antibody that binds to the heterodimer α4β7 integrin and which has shown its efficacy in Ulcerative Colitis (UC) by inducing and maintaining clinical response/remission. The French marketing authorization was obtained for Ulcerative Colitis in patients in failure with anti-Tumor Necrosis Factor (anti-TNF) agents. In the pivotal study, correlation between drug levels and clinical response during induction and maintenance therapy were reported. Moreover, in 3.7% of cases, anti-vedolizumab antibodies were reported during the time-course and 1% had samples that were persistently positive. Up to now, data on the pharmacologic VDZ parameters are scarce and the relationships as well as the predictive value of the measurement of VDZ concentrations and VDZ monoclonal antibodies (mAbs) during the induction and maintenance phases remains unknown. It could be of paramount interest to early identify UC patients under VDZ who will be responders to VDZ induction and to identify those who will achieve clinical remission under maintenance therapy with VDZ.

DETAILED DESCRIPTION:
The contribution of the pharmacokinetic studies of monoclonal antibodies (anti-TNF antibodies currently) has assumed increasing importance of its use in clinical practice. Therapeutic algorithms for both Infliximab (IFX) and Adalimumab (ADA) have been published and are used by many expert teams in the event of loss of therapeutic response. Similarly, the concentrations are assuming important in the indication of therapeutic de-escalation. Lastly, the assays may predict medium-term therapeutic response to treatment and thus enable proposal of preventive therapeutic changes (5). The Gemini 1 study (phase 3 vedolizumab vs. placebo in Ulcerative Colitis) showed a correlation between drug levels and clinical response during induction and maintenance therapy. Moreover, in 3.7% of cases, anti-vedolizumab antibodies were reported during the time-course and 1% had samples that were persistently positive. (1). In addition, we have decided to assess the clinical response to VDZ induction at W10 (Week 10), as the Gemini III trial for Crohn Disease (Crohn Disease) have reported, among patients who had experienced previous Tumor Necrosis Factor (TNF) antagonist failure, that 15% of those given vedolizumab versus 12% under placebo were in remission at W6 (P=0.433) whereas a higher proportion of them were in remission (26%) under VDZ when compared with the placebo arm (12%) at week 10. Therefore, in clinically non-responders at W10, an additional dose of 300 mg of VDZ will be infused at W10 and every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Men or non-pregnant women
* Patients with a diagnosis of ulcerative colitis who requires to start VDZ
* Moderate to severe active ulcerative colitis defined as a total mayo score ranging from 6 to 12 and endoscopic Mayo score above 1
* UC patients with previous failure with TNF antagonist agents and unacceptable side-effects from steroids, and/or immunosuppressive agents (i.e., azathioprine, 6-mercaptopurine, or methotrexate).
* oral prednisone, are allowed at stable dose for at least 4 weeks-before inclusion. Concomitant immunosuppressive agents, mesalamine, are allowed at stable dose for at least three months before inclusion. Steroid tapering has to be set up at Week 6 after starting VDZ, according to the European Crohn's and Colitis Organisation (ECCO) recommendations.
* Informed written consent given.

Exclusion Criteria:

* Existing pregnancy, lactation, or intended pregnancy within the next 15 months
* Minors or History of disease, including mental/emotional disorder that might interfere with their participation in the study
* Serious secondary illnesses of an acute or chronic nature, which in the opinion of the investigator renders the patient unsuitable for inclusion into the study
* Inability to comply with the protocol requirements
* Inability to fill in the diary cards during the last 3 days before each visit
* Severe Acute UC needed hospitalisation
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years)
* Short bowel syndrome
* Previous treatments with vedolizumab, natalizumab, efalizumab or rituximab.
* Previous treatment with adalimumab within 30 days prior enrollment or infliximab and certolizumab pegol within 60 days before enrollment (This period may be shortened in the opinion of the investigator.)
* Prior extensive colonic resection, obstructive (symptomatic) intestinal stricture, abdominal abscess, active or latent tuberculosis,
* Clostridium difficile superinfection;
* Indeterminate colitis
* Concomitant leukocyte apheresis.
* Any contraindication to vedolizumab therapy
* Patients who denied the protocol, not ability to accept or sign consent of the protocol
* Subject involved in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Vedolizumab concentration at week 6 | Week 6
  Determine the optimal threshold of VDZ serum concentration measured at W6 capable to predict the clinical response at week 10 with VDZ.

SECONDARY OUTCOMES:
Vedolizumab concentration at week 14 | Week 14
  Determine the optimal threshold of VDZ serum concentration measured at W14 capable to predict the clinical response at week 52 with VDZ.
vedolizumab concentration and anti-vedolizumab antibodies concentrations at week 2 | Week 2
  Investigating whether the pharmacokinetic parameters of vedolizumab (serum trough levels concentrations, specific antibody concentrations) measured at W2 are predictive of a clinical response and clinical remission at W10.
vedolizumab concentration and anti-vedolizumab antibodies concentrations at week 14 | Week 14
  Investigating whether the pharmacokinetic parameters of vedolizumab (serum trough levels concentrations, specific antibody concentrations) measured at W14 are predictive of a clinical response and clinical remission at W52.
Vedolizumab concentration at week 6 and mucosal healing | Week 6
  Analyzing the value of VDZ trough levels measured at W6 to predict mucosal healing at W10 under induction therapy with VDZ in UC
Vedolizumab concentration at week 14 and mucosal healing | Week 14
  Analyzing the value of VDZ trough levels measured at W14 to predict mucosal healing at W52 under induction therapy with VDZ in UC
intra and inter-individual heterogeneity of VDZ levels | Week 52
  Investigating the intra and inter-individual heterogeneity of VDZ levels within the time-course of VDZ therapy, including the induction and maintenance phases.
Proportion of loss of clinical response | Week 52
  Comparing the proportion of loss of clinical response in responder UC patients as well as in primary non-responders requiring VDZ dose-intensification within one-year of follow-up
Variation of serum VDZ | Week 52
  Assessing the relationships between the variation of serum VDZ trough levels pre- and post-optimization (delta) and the clinical response in primary non-responder patients requiring additional infusions of VDZ.
vedolizumab concentration and anti-vedolizumab antibodies concentrations | Week 52
  Comparing the whole and individual pharmacokinetic parameters (vedolizumab concentration and anti-vedolizumab antibodies concentrations) between patients achieving a clinical remission or not at W52

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ROBLIN, Principal Investigator — CHU SAINT-ETIENNE
Locations (5):
- France (5):
  - CHU Amiens, Amiens
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Chu L'Archet, Nice
  - Ch Lyon Sud, Pierre-Bénite
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No